CLINICAL TRIAL: NCT04688385
Title: IVAC-XS15-CLL01: Personalized Multi-peptide Vaccination in Combination with the TLR1/2 Ligand XS15 in CLL Patients Undergoing Ibrutinib-based Regimes
Brief Title: Personalized Multi-peptide Vaccination in CLL Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iVAC-XS15-CLL01
Record Dates: First submitted 2020-12-08; First posted 2020-12-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: As usual in early phase 1 and 2 studies, statistical planning is designed as such that a statistically reasoned decision for or against a subsequent phase 3 study can be made. The sample size of the study was chosen based on the assumption that, in the case of peptide specific immune response induction in ≤ 30% of the patients, the therapy concept is extended with a probability of at most 5% (type one error, one-sided). On the other hand, in the case of peptide specific immune response induction in ≥ 60% of the patients, the therapy concept should be followed with a probability of at least 80% (power).
  With a sample size of n = 20 patients, this means that at least 10 patients must have an immune response, so that the therapy concept is evaluated in a randomized phase 3 study. The exact power is 87%, the exact type 1 error is 4.8% (calculations based on the binomial distribution with n = 20, p = 0.3 or p = 0.6, k <10 or k ≥ 10).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multipeptide Vaccine + XS 15 (Experimental): a personalizied multi-peptide vaccine in combination with the TLR1/2 ligand XS15 in CLL patients undergoing ibrutinib-based regimes
  Interventions: Biological: Multipeptide Vaccine+ XS15

INTERVENTIONS:
Biological: Multipeptide Vaccine+ XS15 — Peptide vaccination will take place in CLL patients that achieved at least a partial remission with detectable MRD after at least 6 and less than 9 months of an ibrutinib-based treatment regime. MRD will be determined by flow cytometry. MRD positivity is defined as > 10-4 CLL cells in peripheral blood or bone marrow. Patients will receive either ibrutinib monotherapy or combinational therapy before study treatment. Vaccination will be done under ibrutinib monotherapy (i.e. after the end of e.g. anti-CD20 treatment, if applicable).

SUMMARY:
The aim of this study is to evaluate the efficiency along with safety and toxicity of a personalizied multi-peptide vaccine in combination with the TLR1/2 ligand XS15 in CLL patients undergoing ibrutinib-based regimes.

DETAILED DESCRIPTION:
This is a phase I patient-individualized multi-peptide vaccination study in combination with the novel TLR1/2 ligand XS15 in CLL patients under ibrutinib treatment and based on the following rationale:

With the development and clinical success of targeted therapies, the treatment landscape for CLL, which is the most common leukemia in adults, has faced profound changes in the recent years. The disease control achieved by ibrutinib, an inhibitor of the Brutons tyrosine kinase (BTK), has led to its approval as first line therapy. However, in most cases only partial remissions are achieved, and so far perpetual ibrutinib treatment bearing the risk of side effects and development of drug resistance is required. Therefore, current efforts are focusing on the further reduction/elimination of residual CLL cells to allow for reduced treatment time as well as the achievement of long-lasting remissions. A rational and promising approach to achieve this goal is peptide-based immunotherapy, which represents a low side-effect treatment relying on specific immune recognition of tumor-associated HLA presented peptides. Several peptide vaccination studies have reported promising result in terms of in vivo immunogenicity, but so far lacked broad clinical responses. This likely is due to several so far unmet prerequisites for clinical effective peptide vaccination, including the selection of antigens, adjuvants, combinatorial drugs and vaccination time points.

The investigators here adresse these issues as follows:

The reportedly distorted relationship of gene expression and HLA-restricted presentation of the corresponding gene product requires direct methods for peptide target identification for vaccination approaches. This is realized by mass spectrometry-based analysis of the entirety of naturally presented HLA ligands, termed the HLA ligandome of cancer cells. In the recent years, the investigators worked intensively on the characterization of such TAA in HM based on the direct isolation of naturally presented HLA class I and II ligands from leukemia cells and the subsequent identification by mass spectrometry. To allow for the timely and cost-effective production of personalized vaccine cocktail for patients in clinical studies based on HLA ligandome analyses, the investigators have established a so called "warehouse concept" providing premanufactured highly frequent TAA for the formulation of personalized vaccine cocktails. The feasibility of such a warehouse concept, which is utilized in the iVAC-XS15-CLL01 study, was already proven by the investigator's first clinical peptide vaccination study (iVAC-CLL01, NCT02802943). The warehouse has been built based on comprehensive HLA ligandome analysis of CLL cells and composites of a modified cocktail used for the iVAC-CLL01 study as described above. On basis of the individual HLA allotype and a HLA ligandome analysis of CLL cells of the respective patient, 10 tumor-associated peptides are selected from the peptide warehouse. The so-called CLL peptide cocktails (drug substance) are designed to trigger the cellular part of the patients' immune system by activation of CLL-specific T cells. Once activated, these cells can destroy malignant cells presenting the respective antigens. Applying several CLL-associated antigens simultaneously increases the likelihood that a multi-clonal, broad and at the same time highly specific T-cell response is mounted, therebypreventing potential tumor escape mechanisms.

Besides the selection of optimal antigen targets, a further important prerequisite is the use of suitable adjuvant drugs capable to induce potent and long-lasting immune responses. The investigators will use the novel TLR1/2 ligand (XS15, developed in Tübingen) that (i) is water-soluble and (ii) GMP-amenable, (iii) non-toxic and (iv) effective in inducing T cells specific for peptides in vivo.

Another important factor for the clinical effectiveness of peptide-based immunotherapy is the rational combination with standard therapies. In this iVAC-XS15-CLL01 trial, peptide vaccination will be applied in CLL patients under ibrutinib treatment which have achieved at least a partial remission. The remission stage or, even better, the stage of MRD ensures an optimal effector to target cell ratio for peptide-based immunotherapy, as most of the tumor cells are eliminated and the T-cell compartment is recovered. Notably, several studies have proven that ibrutinib does not impair and even can show positive effects on T-cell response.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CLL according to iWCLL guidelines

For Screening phase:

• CLL that warrants treatment (according to modified criteria for initiation of therapy):

* Massive (ie, lower edge of spleen ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly, or
* Massive (ie, ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy, or
* Progressive lymphocytosis in the absence of infection, with an increase in blood ALC ≥ 50% over a 2-month period or lymphocyte doubling time of < 6 months (as long as initial ALC was ≥ 30,000/L), or
* Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy, or -Constitutional symptoms, defined as any one or more of the following disease- related symptoms or signs occurring in the absence of evidence of infection:

  * Unintentional weight loss of ≥ 10% within the previous 6 months, or
  * Significant fatigue (≥ Grade 2), or
  * Fevers > 38.0°C for ≥ 2 weeks, or
  * Night sweats for > 1 month.
* Planned initiation of a ibrutinib-based regime (monotherapy or cominational therapy (e.g. anti-CD20))

For Vaccination phase:

* Ongoing ibrutinib therapy (monotherapy).
* Achievement of a response (at least PR according to iWCLL guidelines)
* MRD positivity (CLL cells in peripheral blood ≥ 10-4, determined by flow cytometry, Labor Kiel, Prof. Brüggemann).
* Negative SARS-CoV-2 test (as long as WHO declares pandemic spread of SARS-CoV-2)
* Prior ibrutinib treatment of at least 6 months and not longer than 8 months.

  * HLA typing positive for any of the following HLA alleles: HLA-A*02, A*24, B*07.
  * Ability to understand and voluntarily sign an informed consent form.
  * Ability to adhere to the study visit schedule and other protocol requirements.
  * Age ≥ 18 years at the time of signing the informed consent form.
  * ECOG performance status score of ≤ 2.
  * Negative serological Hepatitis B test or negative PCR in case of positive serological test without evidence of an active infection, negative testing of Hepatitis C RNA, negative HIV test within 6 weeks prior to study inclusion.
  * Female patients of childbearing potential (FCBP) and male volunteers with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception. This should be started from the signing of the informed consent and continue throughout period of study
  * Postmenopausal or evidence of non-childbearing status. For FCBP: negative urine or serum pregnancy test within 14 days prior to study treatment.

Postmenopausal or evidence of non-childbearing status is defined as:

* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50

Exclusion Criteria:

* Pregnant or lactating females.
* Treatment regimes without ibrutinib
* Ibrutinib-related side effects > CTC grade 2 (CTCAE V5.0)
* Participation in any clinical study or having taken any investigational therapy which would interfere with the study primary and secondary end points.
* Prior history of malignancies other than CLL, unless the subject has been free of the disease for ≥ 5 years. Exceptions include the following:

  * Basal cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Disease transformation (active), i.e. Richter's syndrome, prolymphocytic leukemia.
* Autoimmune hemolysis or immune thrombocytopenia caused by CLL
* Any immunosuppressive treatment not related to CLL except corticosteroids
* Pre-existing auto-immune disease except for Hashimoto thyroiditis and mild (not requiring immunosuppressive treatment) psoriasis
* Chronic lung disease requiring drug treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Induction of a T-cell response after vaccination | Visit 2=Day 30 +/-7days
  60ml of heparin blood for immunomonitoring and analysis of peptide specific T-cell response will be analyzed by the Walz lab, KKE Translational Immunology at the the Department of Immunology, Tübingen (central laboratory). Blood will be taken prior to peptide vaccination on V1, V2, V3, at the end of study visit and the follow up visit.
  Induction of a T-cell response after vaccination on Visit 2, 3, 4 and 5 (follow-up) compared to baseline as determined by IFNγ ELISPOT.
Induction of a T-cell response after vaccination on Visit 3 | Visit 3= Day60 +/- 7days
  60ml of heparin blood for immunomonitoring and analysis of peptide specific T-cell response will be analyzed by the Walz lab, KKE Translational Immunology at the the Department of Immunology, Tübingen (central laboratory). Blood will be taken prior to peptide vaccination on V1, V2, V3, at the end of study visit and the follow up visit.
  Induction of a T-cell response after vaccination on Visit 2, 3, 4 and 5 (follow-up) compared to baseline as determined by IFNγ ELISPOT.
Induction of a T-cell response after vaccination on Visit 4 | Visit 4= 4 to 6 weeks after Visit 3
  60ml of heparin blood for immunomonitoring and analysis of peptide specific T-cell response will be analyzed by the Walz lab, KKE Translational Immunology at the the Department of Immunology, Tübingen (central laboratory). Blood will be taken prior to peptide vaccination on V1, V2, V3, at the end of study visit and the follow up visit.
  Induction of a T-cell response after vaccination on Visit 2, 3, 4 and 5 (follow-up) compared to baseline as determined by IFNγ ELISPOT.
Induction of a T-cell response after vaccination on Visit 5 | Visit 5 =6 months +/- 14 days after Visit 3
  60ml of heparin blood for immunomonitoring and analysis of peptide specific T-cell response will be analyzed by the Walz lab, KKE Translational Immunology at the the Department of Immunology, Tübingen (central laboratory). Blood will be taken prior to peptide vaccination on V1, V2, V3, at the end of study visit and the follow up visit.
  Induction of a T-cell response after vaccination on Visit 2, 3, 4 and 5 (follow-up) compared to baseline as determined by IFNγ ELISPOT.

SECONDARY OUTCOMES:
Immunophenotyping I on Baseline | Baseline
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]
Immunophenotyping I on Visit 1 | Visit 1=Day 1+/-7 days
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]
Immunophenotyping I on Visit 2 | Visit 2=Day 30 +/-7days
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]
Immunophenotyping I on Visit 3 | Visit 3= Day60 +/- 7days
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]
Immunophenotyping I on Visit 4 | Visit 4= 4 to 6 weeks after Visit 3
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]
Immunophenotyping I on Visit 5 | Visit 5 =6 months +/- 14 days after Visit 3
  • Characterization of vaccine induced T-cell responses from Baseline through follow-up: Phenotyping of peptide-specific T-cells by flow cytometry in [%]

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Salih, Prof.Dr., Study Director — CCU Translational Immunology, University Hospital Tuebingen,
Locations (2):
- Germany (2):
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - university Hospital Tuebingen, Tübingen

REFERENCES:
- [Derived] Heitmann JS, Maringer Y, Jung S, Wacker M, Hackenbruch C, Polster M, Marconato M, Nelde A, Bauer J, Zwick M, Baur AS, Lehmann A, Krolla C, Andrieux G, Kohler N, Boerries M, Denk M, Zieschang L, Kammer C, Hoenisch-Gravel N, Richter M, Oezbek MT, Wirths S, Dengler A, Dubbelaar ML, Pumptow M, Martus P, Bruggemann M, Rammensee HG, Salih HR, Walz JS. Personalised multipeptide-based T-cell activator for chronic lymphocytic leukaemia: an open-label, single-centre, phase 1 study. Lancet Haematol. 2026 Jan 14:S2352-3026(25)00323-0. doi: 10.1016/S2352-3026(25)00323-0. Online ahead of print. PMID 41547362
- [Derived] Nelde A, Maringer Y, Bilich T, Salih HR, Roerden M, Heitmann JS, Marcu A, Bauer J, Neidert MC, Denzlinger C, Illerhaus G, Aulitzky WE, Rammensee HG, Walz JS. Immunopeptidomics-Guided Warehouse Design for Peptide-Based Immunotherapy in Chronic Lymphocytic Leukemia. Front Immunol. 2021 Jul 8;12:705974. doi: 10.3389/fimmu.2021.705974. eCollection 2021. PMID 34305947